CLINICAL TRIAL: NCT05598541
Title: Finnish Patient-Reported Outcomes Initiative for Shoulder and Elbow
Acronym: φ-PROMISE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Thomas Ibounig, MD, Helsinki University Central Hospital
Other Study IDs: HUS/715/2021
Record Dates: First submitted 2022-10-26; First posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Cultural Adaptation of Shoulder and Elbow PROMs; Definition of the Patients Acceptable Symptomatic State; Definition of the Minimal Important Difference
Keywords: shoulder; elbow; patient reported outcomes; validation; transcultural adaptation; patients acceptable symptomatic state (PASS); minimal important difference (MID)
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Shoulder: Patients with shoulder problems presenting to the orthopaedic outpatient clinic of the Helsinki University Hospital
  Interventions: Procedure: Surgical or non-surgical treatment
- Elbow: Patients with elbow problems presenting to the orthopaedic outpatient clinic of the Helsinki University Hospital
  Interventions: Procedure: Surgical or non-surgical treatment

INTERVENTIONS:
Procedure: Surgical or non-surgical treatment — Surgical treatment (depending on diagnosis) Non-surgical treatment (such as exercise therapy, pain medication, watch and wait)

SUMMARY:
The purpose of φ-PROMISE project is to carry out a cultural adaptation (translate into Finnish and validate) some of the most frequently used shoulder- and elbow-specific patient-reported outcome measures, PROMs. In addition, we aim to investigate which outcome measures are the most relevant for assessing the severity of complaints and treatment outcomes. Also, we will define the Patients Acceptable Symptomatic State (PASS) and the Minimal Important Difference (MID) of the individual outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Orthopedic outpatient visit at the Helsinki University Hospital
* Signed informed consent
* Age over 18 years
* Finnish as language of communication

Exclusion Criteria:

* Recent surgery (within 2 months)
* Insufficient compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Secondary care outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Validation | 2 weeks
  Assessment of inter- and intra- observer reliability of different outcome measures

SECONDARY OUTCOMES:
PASS | 1 year
  Definition of the Patients Acceptable Symptomatic State for different outcomes
MID | 1 year
  Definition of the Minimal Important Difference for different outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No